CLINICAL TRIAL: NCT07258888
Title: Pulp Transplantation in Necrotic Mature Teeth With Periapical Radiolucency
Acronym: TRANSP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Aliye Kamalak, Assoc Prof, Kahramanmaras Sutcu Imam University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KSU-PT-2024-11; Project No: 2024/3-13D (Other Grant/Funding Number: Scientific Research Projects Coordination Unit of KSU)
Record Dates: First submitted 2025-11-20; First posted 2025-12-02 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Pulpal Regeneration; Pulp Revascularization

STUDY DESIGN:
Intervention Model Description: This study used a parallel-group design with three treatment arms. Twenty-one patients with necrotic mature teeth were randomly assigned (1:1:1 ratio) to one of three groups: Group 1 received autologous dental pulp transplantation, Group 2 received pulp transplantation combined with concentrated growth factor (CGF), and Group 3 underwent conventional root canal therapy. Participants were followed for 12 months to evaluate pulp vitality and periapical healing.
Who Masked: Outcomes Assessor
Masking Description: Outcome evaluations and statistical analyses were performed by blinded examiners independent of the clinical operators.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional Root Canal Therapy (Active Comparator): Patients undergo standard root canal preparation and obturation with gutta-percha and sealer using lateral condensation, followed by restoration.
  Interventions: Procedure: Conventional root canal therapy
- Autologous dental pulp transplantation (Active Comparator): Harvest of autologous third-molar pulp; canal disinfection; transplantation; MTA coronal seal; restoration.
  Interventions: Procedure: Autologous dental pulp transplantation
- Pulp transplantation with CGF (Active Comparator): Same as pulp transplantation with the addition of autologous concentrated growth factor (CGF) placed over the transplanted pulp prior to MTA seal.
  Interventions: Procedure: Pulp transplantation with CGF

INTERVENTIONS:
Procedure: Conventional root canal therapy — Standard root canal instrumentation, irrigation, obturation with gutta-percha and sealer, and restoration.
  Arms: Conventional Root Canal Therapy
Procedure: Autologous dental pulp transplantation — Harvest of autologous pulp tissue from third molar, canal disinfection, placement into recipient tooth, MTA sealing, composite restoration.
  Arms: Autologous dental pulp transplantation
Procedure: Pulp transplantation with CGF — Same as above, but CGF membrane placed over transplanted pulp before MTA sealing.
  Arms: Pulp transplantation with CGF

SUMMARY:
This randomized clinical trial aims to compare autologous dental pulp transplantation alone or combined with concentrated growth factor (CGF) with conventional root canal treatment in necrotic mature teeth with periapical radiolucency. The primary objective is to evaluate whether autologous pulp transplantation can facilitate the return of vitality in necrotic teeth. A secondary objective is to assess whether the addition of CGF provides any further clinical benefit.

Twenty-one patients with single-rooted teeth presenting with periapical lesions are randomly allocated into three groups (n = 7 per group): Group 1 receives autologous pulp transplantation, Group 2 receives pulp transplantation combined with CGF, and Group 3 receives conventional root canal treatment. Donor pulp tissue is obtained from the patient's own non-carious third molars. Clinical and radiographic follow-up is planned at 3, 6, and 12 months, including electrical pulp testing, periapical radiographs, and cone-beam computed tomography (CBCT).

DETAILED DESCRIPTION:
This study investigates the clinical applicability of autologous dental pulp transplantation as a potential biologic treatment alternative for necrotic mature teeth with periapical radiolucency. The trial explores whether transplantation of the patient's own pulp tissue, with or without the addition of concentrated growth factor (CGF), can promote tissue regeneration and functional recovery. The design includes three treatment groups to evaluate the effects of pulp transplantation alone, pulp transplantation combined with CGF, and conventional root canal therapy.

Participants are adults presenting with single-rooted teeth diagnosed with pulp necrosis and periapical pathology. Following randomization, the allocated intervention is performed under standardized clinical protocols. Donor pulp tissue is harvested atraumatically from non-carious third molars of the same patient. Outcome assessments include vitality testing and radiographic evaluations at predetermined follow-up intervals. The study aims to provide foundational clinical evidence regarding the feasibility, safety, and regenerative potential of autologous pulp transplantation techniques to inform future clinical applications.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-40 years
* Presence of single-rooted permanent teeth diagnosed with:
* Pulp necrosis or
* Irreversible pulpitis with radiographic periapical lesions
* Availability of a caries-free, periodontally healthy third molar suitable for donor pulp harvesting

Good general health, with no systemic diseases

-Ability to understand the study procedures and provide written informed consent

Exclusion Criteria:

* Multi-rooted teeth or teeth with complex canal anatomy
* Systemic diseases or medical conditions that may affect wound healing (e.g., diabetes, immunosuppression)
* Lack of a suitable donor third molar for pulp harvesting
* Advanced periodontal attachment loss or active periodontal disease
* Pregnancy or lactation
* Recent use of antibiotics or anti-inflammatory drugs (<1 month)
* Inability or unwillingness to attend scheduled follow-ups

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2023-11-05 (Actual); Primary Completion 2023-11-05 (Actual); Study Completion 2025-09-05 (Actual)

PRIMARY OUTCOMES:
Pulp Vitality Recovery Assessed by Electric Pulp Test | 12 months after treatment
  Assessment of the percentage of treated teeth exhibiting a positive response to the Electric Pulp Test, indicating return of pulp vitality (revascularization or functional regeneration).
  Unit of Measure:
  % of teeth with positive EPT response
  Measurement Tool:
  Electric Pulp Test (EPT)

SECONDARY OUTCOMES:
Adverse Events Related to Transplantation Procedures | Throughout 12-month follow-up period
  Incidence of postoperative pain, swelling, infection, or any other adverse event following treatment.
  Unit of Measure:
  % of participants experiencing any adverse event
  Measurement Tool:
  Clinical examination and patient-reported symptom assessment
Pulp Vitality Recovery | 12 months after treatment
  Return of pulp vitality assessed by an electric pulp test (EPT). A positive response to EPT indicates revascularization or functional pulp regeneration after treatment.
  Unit of Measure:
  % of teeth with positive EPT response
  Measurement Tool:
  Electric Pulp Test (EPT)

CONTACTS AND LOCATIONS:
Overall Officials: Aliye Kamalak, Associate Professor Dr., Principal Investigator — Kahramanmaraş Sütçü İmam University, Faculty of Dentistry, Department of Endodontics
Locations (1):
- ahramanmaraş Sütçü İmam University, Faculty of Dentistry, Kahramanmaraş, onikişubat, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) that support the findings of this study will be available from the corresponding author upon reasonable request after publication. Data will include anonymized clinical outcomes and statistical analysis files, excluding any information that could compromise participant privacy.
Supporting Information: Study Protocol, SAP
Time Frame: De-identified individual participant data and supporting documents will be available beginning 9 months after publication of the study results, with no fixed end date for data availability.
Access Criteria: Access will be granted to qualified researchers upon reasonable written request to the corresponding author (aliyekamalak@gmail.com). Requesters must provide a brief research proposal and obtain approval from the Institutional Ethics Committee. Data will be shared electronically in anonymized form.

REFERENCES:
- [Result] Cehreli ZC, Unverdi GE, Ballikaya E. Deciduous Tooth Pulp Autotransplantation for the Regenerative Endodontic Treatment of Permanent Teeth With Pulp Necrosis: A Case Series. J Endod. 2022 May;48(5):669-674. doi: 10.1016/j.joen.2022.01.015. Epub 2022 Feb 1. PMID 35114270
- [Result] Yan H, De Deus G, Kristoffersen IM, Wiig E, Reseland JE, Johnsen GF, Silva EJNL, Haugen HJ. Regenerative Endodontics by Cell Homing: A Review of Recent Clinical trials. J Endod. 2023 Jan;49(1):4-17. doi: 10.1016/j.joen.2022.09.008. Epub 2022 Oct 18. PMID 36270575
- [Result] Kim U, Kim S, Choi SM, Kang MK, Chang I, Kim E. Regenerative Endodontic Procedures With Minced Pulp Tissue Graft in Mature Permanent Teeth: A Clinical Study. J Endod. 2025 Jan;51(1):43-53.e2. doi: 10.1016/j.joen.2024.10.004. Epub 2024 Oct 12. PMID 39401572
- See also: Official website of the Faculty of Dentistry, Kahramanmaraş Sütçü İmam University - the institution where the study was conducted. — https://dishekimligi.ksu.edu.tr/
- Available data/document: Individual Participant Data Set — https://dishekimligi.ksu.edu.tr/ — Data sharing will follow institutional policies and ethical guidelines to ensure participant confidentiality.